CLINICAL TRIAL: NCT04424732
Title: Stereotactic Body Radiotherapy for Bone Only Oligometastatic Breast Cancer: A Prospective Study
Brief Title: SBRT for Breast Cancer Oligometastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Abdulmajeed Dayyat, Consultant Radiation Oncologist, King Hussein Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20 KHCC 91
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Breast Neoplasm Malignant Female
Keywords: Stereotactic Body Radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiotherapy for Breast Bony oligometastases (Other): Newly diagnosed bone only oligometastatic breast cancers with 1-3 bone metastases will be enrolled in this protocol. Patients will receive SBRT to all metastatic sites.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — This is a prospective study of breast bone only oligometastases (up to three sites). Following systemic treatment and primary tumor control, patients will receive SBRT to all metastatic sites. Data on toxicities and oncological outcomes will be collected for future analysis. There will be no change in the standard systemic therapy nor the local therapy of the primary tumor.

SUMMARY:
This is a prospective data collection of treatment outcome for newly diagnosed oligometastatic breast cancers with 1-3 bone metastases. Eligible patients will be identified from the weekly Breast MDC. Patients will receive the recommended systemic and local treatment (including metastases directed SBRT) according to our clinical practice guidelines.Patients will be followed according to our routine with clinical and radiologic assessment. It is preferred that the same imaging method that was used to originally detect the metastases be used in follow-up assessments. The first imaging for SBRT sites will be three months post SBRT and every three months for the first year, every 6 months for the second year, then annually. Response and progression for these metastases will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions is used in the RECIST criteria. If functional imaging (bone scan, PET) were used at staging, changes in the uptake will be used in follow up scans to determine response to treatment and progression. As for SBRT related morbidities, we will use the Common Terminology Criteria for Adverse Events (CTCAE v5) for toxicity reporting and scoring.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years old with a pathologically proven breast cancer who present with 1-3 bone metastases will be included.
* Metastases need to be confirmed pathologically if possible, otherwise two different imaging modalities (CTor MRI and bone scan or PET) are needed to confirm metastases.
* Patients should be able to receive the recommended local and systemic treatment and the primary tumor must be controlled at time of SBRT.
* Maximum diameter of individual metastasis metastasis in any dimension ≤ 5 cm; and must be >5 cm away from each other (defined as Edge to Edge of tumor).

Exclusion Criteria:

* Non bone metastatic breast cancers
* Prior history of radiotherapy to same sites of SBRT
* Pathologic fractures of involved bones
* Contraindications to radiotherapy including pregnancy and connective tissue disease.
* Patients with impaired cognitive functions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 5 years
  the interval from diagnosis until disease progression
Overall survival (OS) | 5 years
  time from diagnosis to death from any cause or last follow-up

SECONDARY OUTCOMES:
Existing metastasis control | 3 years
  the interval from diagnosis until local progression of the treated metastases
Appearance of new metastases | 3 years
  the interval from diagnosis until appearance of new metastases
Adverse Events | 3 years
  CTCAE v5. for acute and chronic toxicity reporting and scoring

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmajeed Dayyat, MD, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Jordan